# **Protocol information**

# **Full title:**

Impulse Oscillometry Measurements in Severe Eosinophilic Asthmatics Before and After Anti-IL-5 Factor Initiation (IMPOSE)

**ClinicalTrials.gov ID NCT05147155** 

**Sponsor** University of Thessaly

Information provided by Ourania Kotsiou, University of Thessaly (Responsible Party)

Last Update Posted 2024-05-10

## Title of the trial for lay people, in easily understood, i.e., non-technical, language:

Impulse oscillometry as a method to document and monitor the efficacy of anti-IL-5 factor in patients with severe eosinophilic asthma.

#### **SCIENTIFIC RATIONALE**

Asthma is an inflammatory airways disease affecting the entire bronchial tree. The importance of small airways in asthma has been well documented [1,2]. Small airways defined as those with an internal diameter of 2 mm or less, which referred to as the silent zone of the lungs. Small airway disease (SAD) is present across patients with all stages of asthma, but it is particularly prevalent in those with more severe disease and more frequent symptoms [3]. Particularly, the silent zone has been related to asthma control, severity, and risk of exacerbation [3,4]. SAD is more prevalent in asthmatic patients with fixed airflow obstruction compared to asthmatic patients without fixed airflow obstruction [5].

The small airways contribute to the resistance in the airways of patients with obstructive airways disease [6]. It was estimated that total small airways resistance was 24% of total airway resistance in healthy adults and increased to 34% in asymptomatic newly diagnosed patients with asthma and 51% in patients with severe asthma [4].

Structural alterations at the peribronchiolar level contribute to the pathogenesis of functional abnormalities observed in patients with severe asthma [7]. Remodeling can affect small airway wall stiffness, thereby changing their distensibility [8]. An increase in type collagen, matrix metalloproteinase and fibronectin and a decrease in collagen III localized to the outer part of the lung were found in patients who died of asthma [9]. It has been recently documented that those structural abnormalities in patients with severe asthma associated with a higher frequency of exacerbations, worse asthma severity, quality of life, and asthma control [3]. Moreover, it has been reported reproducibly higher alveolar NO concentrations in refractory asthma group compared to mild-moderate asthma group, supporting the hypothesis that refractory asthma is associated with distal lung inflammation [10].

Although it is increasingly recognized that the small airways play an important role in severe asthma and SAD may complicate severe asthma treatment, it is notoriously difficult to measure small airways inflammation and/or dysfunction [11,12]. SAD is a complex and silent signature of severe asthma that is likely to be directly or indirectly captured by combinations of physiological tests, such as spirometry, body plethysmography, impulse oscillometry (IOS), and multiple breath nitrogen washout. For clinical practice, it is important to adopt easy-to-use clinical measures, such as IOS and spirometry, to delineate various severe asthma SAD subtypes.

Heterogeneous airway narrowing is a significant marker of severe asthma related to resistance and reactance [13]. IOS seemed to have better sensitivity to detect SAD than effort-dependent forced expiratory flow between 25% and 75% (FEF25-75%) [11]. Spirometry, which is the standard method for measurement of pulmonary function, is unlikely to reflect the pathophysiology of SAD since it measures bulk flow propagating predominantly from the larger central airways; therefore, there are limitations in detecting changes in small airways and airway trapping in patients with asthma [14]. Furthermore, spirometry performance remains challenging for many elderly patients who have comorbidities that affect the test procedure, as well as in cases where patient cooperation is lacking, such as children or patients with physical and cognitive limitations [14]. Therefore, a more readily available test for SAD is crucial for patient assessment.

The use of commercialized forced oscillation technique (FOT) devices to assess impedance in obstructive diseases such as asthma has gained popularity. The earlier FOT instruments allowed only one sound frequency to be passed at a time. Some of the more recent FOTs now use sound waves of two or three different frequencies at one time [15]. IOS is an improvised technique of that FOT that could use multiple sound frequencies at one time [16]. Although FOT devices are generally comparable, IOS is the most commonly used type of FOT in clinical practice [17]. IOS is a noninvasive and convenient technique to measure both airway resistance and reactance during tidal breathing by an effort-independent and patient-friendly modality for evaluating lung function and peripheral airway dysfunction [18], providing extensive description of oscillatory pressure and giving better mathematical analyses of resistance and reactance using the fast Fourier transform (FFT) technique compared to FOT. In FOT, the sound waves of different frequencies were transmitted sequentially, whereas in IOS, an impulse, which can be mathematically decomposed into different frequencies, is transmitted. This helps in reducing the time of the test and also provides a high signal to noise resolution [18]. Resistance can be conceptualized as a sound wave requires to travel through the airways and inflate the lung [19]. The reactance of the respiratory system is composed of the inert and elastic properties of the respiratory system. The sum of the forces ahead of the sound wave (resistance) and those generated behind the sound wave in response to the pressure of the wave (reactance) equal the impedance of the entire respiratory system; thus permits passive measurement of lung mechanics [19]. Importantly, IOS can differentiate small airway obstruction from large airway obstruction and is more sensitive than spirometry for peripheral airway disease [13,19].

The clinical classification of SAD into subtypes by use of IOS is meaningful, given its association with GINA severity stages, asthma control, quality of life, and exacerbations. IOS can be useful in determining baseline lung function, demonstrating a response to bronchodilator or bronchoprovocation, and predicting asthma exacerbations and loss of disease control especially, in children and elderly with

obstructive airway diseases [20]. Moreover, the SAD subtype classification with IOS has been used to determine the inhaled corticosteroids particle size is needed for proper airway inflammation treatment [21].

Eosinophilic inflammation in the small airways of patients with severe asthma is considered to be an important marker of disease severity [2,22,23). In clinical trials, treatment with mepolizumab reduces exacerbation rates by almost a half along with modest improvements in symptom scores and forced expiratory volume in 1 s (FEV $_1$ ) early after the first month of commencing mepolizumab treatment [23,24]. However, there is an apparent discrepancy between major patient-reported outcomes and lung function that should be explored.

It has recently been reported that mepolizumab improves small airway function in severe eosinophilic asthma as detected by multiple-breath nitrogen washout test [23]. The improvement in small airway function was seen rapidly after the first mepolizumab injection and was associated with a sustained response in the majority of patients [23]. However, gaps in knowledge about the choice of device, gas, and standardization across systems are key issues leading the committee to conclude that multiple-breath nitrogen washout test is not ready for use as a clinical trial endpoint in asthmatics [16].

In the past few months, Antonicello et al. provided data showed that FOT could be an effective method to document and monitor the efficacy of mepolizumab in treating severe eosinophilic asthma. In this study, FOT detected early treatment-induced changes in peripheral airways function [25]. This study included 18 patients with severe eosinophilic asthma, candidates for mepolizumab therapy, and no other control groups were enrolled [25]. These preliminary results motivate further prospective studies to evaluate respiratory mechanics using other FOT devices such as the IOS; thus enriching the knowledge regarding the small airway asthma phenotype by unlocking the lung's quiet zone.

#### **HYPOTHESIS**

We hypothesize that early improvement in small airway function may be a significant contributor to the therapeutic response of anti-IL-5 monoclonal antibody therapy in patients with severe uncontrolled eosinophilic asthma. We speculate that SAD could be effectively evaluated using IOS. Consequently, this study could lead to novel SAD subtypes with possible clinical relevance in the context of treatment with anti-IL-5 factor. We hypothesize that healthy individuals and patients with severe controlled asthma would disclose a lesser extent of SAD than patients with severe uncontrolled eosinophilic asthma with or without fixed airway obstruction.

#### **OBJECTIVES**

We sought to describe early changes in respiratory mechanics by means of IOS in patients with severe eosinophilic asthma commencing mepolizumab treatment. The detected parameters will be compared to a group of matched for age and gender healthy controls as well as with a group of patients with severe controlled asthma matched for age and gender requiring high dose inhaled corticosteroids (ICS) /long-acting beta-agonist (LABA) combination therapy to prevent asthma from becoming uncontrolled.

#### **METHODS**

### **Study Population**

Our sample will consist of 40 patients between 18 and 82 years of age with uncontrolled severe eosinophilic asthma despite receiving high dose ICS/LABA combination therapy.

## Principal inclusion criteria:

- Written informed consent
- Male or female outpatient aged 18 to 82 years inclusive
- History of bronchial asthma for at least six months as defined by ATS criteria
   [26].
  - The patients will be required to have one or more of the following objective physiological criteria: positive results on methacholine or mannitol challenge during the previous year, bronchodilator reversibility to 400 mg of inhaled Salbutamol of FEV<sub>1</sub>  $\geq$ 12% and 200ml or peak flow variability of  $\geq$ 20% over two weeks.
- Diagnosis of severe asthma, defined as asthma that requires treatment with high dose inhaled corticosteroids plus a second controller and/or systemic corticosteroids to prevent it from becoming uncontrolled or that remains uncontrolled despite this therapy [27, 28].
  - All patients will be medicated with at least 880  $\mu$ g of fluticasone propionate or the equivalent by inhalation per day and at least three months of treatment with an additional controller. Patients will be allowed to continue their antiasthma therapy throughout the study.
- Patients should have uncontrolled asthma commencing mepolizumab treatment, based on investigator assessment, including one or both of the following:

- -Poor symptom control (frequent symptoms or reliever use, activity limited by asthma, night waking due to asthma), defined as ACQ consistently  $\geqslant$ 1.5 or ACT<20.
- -Frequent exacerbations ( $\geq 2$ /year) requiring oral corticosteroids, or severe exacerbations ( $\geq 1$ /year) requiring hospitalization or burst of systemic corticosteroids ( $\geq 3$  days) [29].
- All patients will have an eosinophil count of at least 150 cells per microliter in the peripheral blood at screening or at least 300 cells per microliter at some time during the previous year.

## **Control groups**

Control groups will be a set of 50 healthy individuals matched for age and gender and 40 patients with severe well-controlled asthma requiring high dose ICS/LABA combination therapy from becoming uncontrolled, as previously defined, matched for age and gender.

#### Principal exclusion criteria:

- Diseases and health status:
  - -clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation
  - -suffering from COPD (i.e., chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
- Asthmatic patients and healthy controls currently smoking or with a smoking pack history greater than 10 will be excluded.

#### Common exclusion criteria:

- pregnancy
  - -intention to become pregnant during the course of the study
  - -breast feeding
  - -participation in another study within the 30 days preceding and during the present study
  - -known or suspected non-compliance, alcohol or drug abuse
  - -inability to follow the procedures of the study, e.g., due to language problems, psychological disorders

## Sampling

Approximately 1000 patients with asthma per year are treated in the external Unit of Asthma of Respiratory Medicine Department of the University of Thessaly in

Greece. Nevertheless, in order to certainly achieve the estimated study sample size, to maximize the response rate and to reduce survey error, the Respiratory Medicine Department of the University of Thessaly will cooperate with a network of private respiratory physicians in Central and Northern Greece that serves a population base of about 3,000,000. Asthma education programs will regularly take place to raise severe asthma awareness, improve asthma control and management by creating a community Interlink between Respiratory Medicine Department and private sector from across central and northern Greece.

Furthermore, Respiratory Medicine Department of the University of Thessaly, via more than 12 clinical-community partnership spirometry surveillance programs with ten primary Health Care Centers in Central and Northern Greece, has already created a network of researchers, experts, and healthcare practitioners which is vitally important to early identify patients with uncontrolled asthma.

#### **Ethics**

Verbal and written informed consent will be obtained from all subjects before the study, according to the Helsinki declaration [30]. The protocol has already been approved by the Larissa University Hospital Ethics Committee (Approval number: 48841/25/10/2019)

**Target enrolment/sample size:** (Required for clinical studies)

130 (40 patients with severe uncontrolled eosinophilic asthma commencing mepolizumab treatment, 40 patients with severe controlled asthma medicating with high dose ICS/LABA combination therapy, and 50 healthy individuals matched for age and gender)

Anticipated rate of enrolment: (Required for clinical studies)

1 to 4 patients per month

Estimated study start date: (FSFV/Study Start/Analysis Start)
May 2020

Estimated study completion date: (LSLV/Study End/Analysis Complete)
September 2023

## **Study Design and Methods**

This will be a 2-year prospective, cohort study. Patients will receive mepolizumab, which will be administered as a 100-mg subcutaneous dose every four weeks. Subjects

will be present for subcutaneous mepolizumab (100 mg) injection initially at visit 0 (Week 0), then for reassessment at two (Week 2) and four weeks (Week 4) and continued monthly treatment with reassessment at three (Week 12) and six months (Week 26). The patients will not alter their usual treatment regimen between Week 0 and Week 12; thus mitigating any other potential confounder.



Detailed lung function tests will be performed at visit 0 in the following order: the fraction of exhaled nitric oxide (FeNO), IOS performance then spirometry and lung volumes measurement. All testing will be conducted before and 30 minutes after mepolizumab injection. Asthma control and quality of life questionnaires will be filled. All testing will be conducted on Week 0, Week 4, Week 12 and Week 26.

#### Measurements

At each clinic visit, we will evaluate the results of spirometric, IOS and lung volumes tests and will administer the 5-item Asthma Control Questionnaire (ACQ-5), Asthma Control Test (ACT), and Asthma Quality of Life Questionnaire (AQLQ).

#### Asthma control questionnaire (ACQ-5)

Symptom control will be determined using the symptom-only 5-item asthma control questionnaire (ACQ-5). A score > 1.5 indicates poor control and an individual change > 0.5 is clinically important [31].

## Asthma Control Test (ACT)

The ACT will provide us with a snapshot of how well asthma has been controlled over the last four weeks, giving a score out of 25. A score of less than 20 means that asthma may not have been controlled during the past four weeks [32].

#### Asthma Quality of Life Questionnaire (AQLQ)

The Asthma Quality of Life Questionnaire (AQLQ) is a 20-item self-administered questionnaire that covers four dimensions (breathlessness, mood, social limitation and worrying) and gives a total score and subscales scores. Patients have to respond to a series of statements describing how asthma (or its treatment) affects them and indicate which option closely applies to them over the past four weeks. A score of 10 corresponds to a maximum impairment of quality of life and a score of 0 corresponds to no impairment [33].

## **Lung function tests**

# Fraction of exhaled nitric oxide (FeNO).

The fraction of exhaled nitric oxide (FeNO) (MEDISOFT, MEDICAL GRAPHICS CORP, Minnesota, USA) will be performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines [20]. Recommended cutoff values for normal FeNO levels < 25 parts per billion (ppb) and elevated FeNO > 50 ppb have been published [34,35].

### Impulse Oscillometry (IOS)

IOS measurements will be performed in triplicate according to standard guidelines, with a Jaeger MasterScreen IOS system (Carefusion, Germany, JLAB software version 5.22.1.50) [36-38]. A volume calibration will be performed daily using a 3-L volume syringe, and the accuracy of resistance measurements will be confirmed daily using a standard 0.2 Kpa.s.L<sup>-1</sup> resistance mesh. Each patient will be seated upright, wear a nose clip, and press on their cheeks with their hands to prevent an upper airway shunt. To avoid air leakage, patients will seal their lips tightly around the mouthpiece [39-41]. While the impulse will be produced by the speaker is moving with the patient's breathing, a pressure and flow transducer will be measure inspiratory and expiratory flow and pressure changes in the respiratory system. Mean values for resistance at 5 Hz (R5: indicates total airway resistance); resistance at 20 Hz (R20: approximates central airway resistance); the difference between R5 and R20 (R5-R20: considered to be an index for small airways); reactance at 5 Hz (X5: relates to compliance); resonant frequency (Fres); and integrated area of low-frequency X (AX) values will be derived as previously reported [41-44]. Fres and AX are values that detect expiratory flow limitations. R5-R20 and AX are thought to reflect changes in the quiet zone of the lungs [45]. IOS data will be carefully reviewed offline and qualityassured by professor K.I Gourgoulianis, an expert clinician, to reject segments affected by airflow leak or swallowing artifacts. Acceptability criteria for IOS measurements will include coherence values of ≥0.6 at 5 Hz, between test coefficient of variation of Zrs of <15% (with a minimum of three tests) and the absence of the following features within the flow tracings gauged by visual inspections (swallowing, glottis closure, leak around the mouthpiece, improper seal with the nose clip). The best of three acceptable attempts with the lowest respiratory resistances will be chosen for the final data analysis. During this study, one technician will obtain all IOS measurements.

Prof. Gourgoulianis make substantial contributions to the clinical application of airway diseases with more than 300 publications in this research area [46-68], performing measurements with FOT over several decades, be able to educate a number of respiratory physicians in Respiratory Medicine Department of University of Thessaly by sharing his vast expert knowledge in pulmonary physiology, FOT, and IOS testing and related areas.

## **Spirometry**

Spirometry (Spirolab, MIR, Rome, Italy) will be performed according to ATS/ERS guidelines [69]. Predicted values will be derived from the Global Lung Initiative [70]. To avoid any negative effects of forced expiration on the airway, spirometry will never be performed before the IOS measurements. The percent predicted forced vital capacity (%FVC), the percent predicted forced expiratory volume in 1 s (%FEV<sub>1</sub>), the FEV<sub>1</sub>/FVC ratio, the percent predicted the maximal mid-expiratory flow (%MMEF), and the percent predicted peak expiratory flow (%PEF) would be obtained. The best of at least three technically acceptable results will be selected.

## Constant volume plethysmograph

Lung volumes measurement [total lung capacity (TLC), residual volume (RV), ratio of RV/TLC], and airway resistance (Raw) will be measured in a constant volume plethysmograph (CardinalHealth, Yorba Linda, CA, USA) as previously described [71,72].

## **Study Endpoints**

### The study endpoints will be:

1) To describe early and late changes in respiratory mechanics by means of IOS in patients with severe eosinophilic asthma commencing mepolizumab treatment.

### The secondary study endpoints will be:

- 1) To identify differences in respiratory mechanics by means of IOS in patients with severe uncontrolled eosinophilic asthma prior to anti-IL-5 therapy compared to healthy individuals.
- To identify differences in respiratory mechanics by means of IOS in patients with severe eosinophilic asthma commencing anti-IL-5 treatment compared to patients with severe controlled asthma medicated high dose ICS/LABA combination therapy.
- 3) To investigate the association between RV/TLC ratio, FeNO, spirometric values and IOS measurements in patients with severe uncontrolled asthma before and after mepolizumab treatment.
- 4) To investigate the association between the changes in respiratory mechanics by means of IOS and asthma control measurement as defined by ACT and ACQ-

- 5 questionnaires in patients with severe eosinophilic asthma before and after mepolizumab treatment.
- 5) To investigate the association between the changes in respiratory mechanics by means of IOS and the quality of life measurement as defined by AQLQ in patients with severe eosinophilic asthma before and after mepolizumab treatment.

#### **Statistical Plan or Data analysis**

Data will be analyzed using the statistical program SPSS 22 (IBM Corporation, Armonk, NY, USA). Quantitative variables will be presented as mean with standard deviation (SD), and qualitative variables will be presented as frequencies with percentages. Chisquare test will be used to explore any associations between qualitative variables. To identify differences between two independent groups when the dependent variable will either ordinal or continuous, unpaired t-tests or Mann–Whitney U tests will be used for normally distributed and skewed data, respectively. Differences between more than two unrelated groups will be tested by one-way analysis of variance (ANOVA). A result will be considered statistically significant when the P-value will be <0.05.

## Limitations

This will be the first study to investigate small airway dysfunction using IOS in patients with severe uncontrolled eosinophilic asthma commencing mepolizumab treatment. While oscillometry measurements are portrayed as a marker of small airway dysfunction, the normal reference ranges or threshold to define SAD has not been established yet. However, IOS has many advantages as is the most commonly used type of FOT in clinical practice including the use of simple tidal breathing maneuvers against forced maneuvers applied in spirometry and thus require less effort, while it demonstrates a change in early disease wherein spirometry is normal [16].

# What is your planned publication? Abstract, Manuscript, Study report

- Planned Publication date (Abstract):
   January 2022
- Planned Publication date (Manuscript):

## March 2022

Planned Publication Date (Study report):
 March 2020

| Planned Publication Date (Study report) | Planned Publication date (Abstract) | Planned Publication date (Manuscript) |
|---|---|---|
| March 2020 | January 2022 | March 2022 |

# References

- 1. Farah CS, King GG, Brown NJ, Peters MJ, Berend N, Salome CM. Ventilation heterogeneity predicts asthma control in adults following inhaled corticosteroid dose titration. J Allergy Clin Immunol. 2012;130:61–8.
- 2. Kraft M, Pak J, Martin RJ, Kaminsky D, Irvin CG. Distal lung dysfunction at night in nocturnal asthma. Am J Respir Crit Care Med. 2001;163:1551–6.
- 3. Postma DS, Brightling C, Baldi S, Van den Berge M, Fabbri LM, Gagnatelli A, Papi A, Van der Molen T, Rabe KF, Siddiqui S, Singh D, Nicolini G, Kraft M, ATLANTIS study group. Exploring the relevance and extent of small airways

- dysfunction in asthma (ATLANTIS): baseline data from a prospective cohort study. Lancet Respir Med.2019;7:402-16.
- 4. Carr TF, Altisheh R, Zitt M. Small airways disease and severe asthma. World Allergy Organ J. 2017;10:20.
- 5. Pornsuriyasak P, Khiawwan S, Rattanasiri S, Unwanatham N, Petnak T. Prevalence of small airways dysfunction in asthma with- and without-fixed airflow obstruction and chronic obstructive pulmonary disease. Asian Pac J Allergy Immunol. 2019 Jun 4.
- 6. Van der Wiel E, ten Hacken NH, Postma DS, van den Berge M. Small-airways dysfunction associates with respiratory symptoms and clinical features of asthma: a systematic review. J Allergy Clin Immunol. 2013;131:646–57.
- 7. Mauad T, Silva LF, Santos MA, Grinberg L, Bernardi FD, Martins MA, Saldiva PH, Dolhnikoff M. Abnormal alveolar attachments with decreased elastic fiber content in distal lung in fatal asthma. Am J Respir Crit Care Med. 2004;170:857-62.
- 8. Nihlberg K, Andersson-Sjöland A, Tufvesson E, Erjefält JS, Bjermer L, Westergren-Thorsson G. Altered matrix production in the distal airways of individuals with asthma. Thorax. 2010;65:670–76.
- 9. Dolhnikoff M, da Silva LF, de Araujo BB, Gomes HA, Fernezlian S, Mulder A, Lindeman JH, Mauad T. The outer wall of small airways is a major site of remodeling in fatal asthma. J Allergy Clin Immunol. 2009123:1090-7.
- 10. Berry MA, Shaw DE, Green RH, Brightling CE, Wardlaw AJ, Pavord ID. The use of exhaled nitric oxide concentration to identify eosinophilic airway inflammation: an observational study in adults with asthma. Clin Exp Allergy. 2005;35:1175-9.
- 11. van den Berge M, Kerstjens HAM. Finally More Direct Evidence that Impulse Oscillometry Measures Small Airways Disease. Am J Respir Crit Care Med. 2019 Jun 12.
- 12. van der Wiel E, Postma DS, van der Molen T, Schiphof-Godart L, Ten Hacken NH, van den Berge M. Effects of small airway dysfunction on the clinical expression of asthma: a focus on asthma symptoms and bronchial hyperresponsiveness. Allergy. 2014;69:1681-8.
- 13. Bhatawadekar SA, Leary D, Maksym GN. Modelling resistance and reactance with heterogeneous airway narrowing in mild to severe asthma. Can J Physiol Pharmacol. 2015;93:207-14.
- 14. Park JH, Lee JH, Kim HJ, Jeong N, Jang HJ, Kim HK, Park CS. Usefulness of impulse oscillometry for the assessment of bronchodilator response in elderly patients with chronic obstructive airway disease. J Thorac Dis. 2019;11:1485-94.

- 15. Brashier B, Salvi S. Measuring lung function using sound waves: role of the forced oscillation technique and impulse oscillometry system. Breathe (Sheff). 2015;11:57-65.
- 16. Desai U, Joshi JM. Impulse oscillometry. Adv Respir Med. 2019;87:235-8.
- 17. Soares M, Richardson M, Thorpe J, Owers-Bradley J, Siddiqui S. Comparison of Forced and Impulse Oscillometry Measurements: A Clinical Population and Printed Airway Model Study. Sci Rep. 2019;9:2130.
- 18. Bickel S, Popler J, Lesnick B, Eid N. Impulse oscillometry: interpretation and practical applications. Chest. 2014;146:841-7.
- 19. Smith HJ, Reinhold P, Goldman MD. Forced Oscillation Technique and Impulse Oscillometry. Lung Function Testing: European Respiratory Society Monograph. Sheffield (England): European Respiratory Society; 2005. p. 72–105.
- 20. McDowell KM. Recent Diagnosis Techniques in Pediatric Asthma: Impulse Oscillometry in Preschool Asthma and Use of Exhaled Nitric Oxide. Immunol Allergy Clin North Am. 2019;39:205-19.
- 21. Sugawara H, Saito A, Yokoyama S, Tsunematsu K, Takahashi H. Comparison of therapeutic effects of inhaled corticosteroids on three subtypes of cough variant asthma as classified by the impulse oscillometry system. Respir Res. 2019;20:41.
- 22. Carroll N, Cooke C, James A. The distribution of eosinophils and lymphocytes in the large and small airways of asthmatics. Eur Respir J. 1997;10:292–300.
- 23. Farah CS, Badal T, Reed N, Rogers PG, King GG, Thamrin C, Peters MJ, Seccombe LM. Mepolizumab improves small airway function in severe eosinophilic asthma. Respir Med. 2019;148:49-53.
- 24. Ortega HG, Liu MC, Pavord ID, Brusselle GG, FitzGerald JM, Chetta A, Humbert M, Katz LE, Keene ON, Yancey SW, Chanez P. For the MENSA Investigators. Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2014;371:1198–207.
- 25. Antonicelli L, Tontini C, Marchionni A, Lucchetti B, Garritani MS, Bilò MB. Forced oscillation technique as method to document and monitor the efficacy of mepolizumab in treating severe eosinophilic asthma. Allergy. 2019 Jun 5. doi: 10.1111/all.13938.
- 26. Aaron SD, Boulet LP, Reddel HK, Gershon AS. Underdiagnosis and Overdiagnosis of Asthma. Am J Respir Crit Care Med. 2018;198:1012-20.
- 27. Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014;43:343-73.

- 28. "International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma." Kian Fan Chung, Sally E. Wenzel, Jan L. Brozek, Andrew Bush, Mario Castro, Peter J. Sterk, Ian M. Adcock, Eric D. Bateman, Elisabeth H. Bel, Eugene R. Bleecker, Louis-Philippe Boulet, Christopher Brightling, Pascal Chanez, Sven-Erik Dahlen, Ratko Djukanovic, Urs Frey, Mina Gaga, Peter Gibson, Qutayba Hamid, Nizar N. Jajour, Thais Mauad, Ronald L. Sorkness and W. Gerald Teague. Eur Respir J. 2018;52. pii: 1352020.
- 29. Global Initiative for Asthma, 2018. Available from: https://ginasthma.org/wp-content/uploads/2018/11/GINA-SA-FINAL-wms.pdf
- 30. Yu M, Fischhoff B, Krishnamurti T. Implementing a New Common Rule Requirement for Informed Consent: A Randomized Trial on Adult Asthma Patients. MDM Policy Pract. 2019;4:2381468319839315.
- 31. Juniper EF, Svensson K, Mork AC, Stahl E. Measurement properties and interpretation of three shortened versions of the asthma control questionnaire. Respir Med. 2005;99:553–8.
- 32. Sonia Cajigal, Karen E. Wells, Edward L. Peterson, Brian K. Ahmedani, James J. Yang, Rajesh Kumar, Esteban G. Burchard, L. Keoki Williams. .Predictive properties of the Asthma Control Test and its component questions for severe asthma exacerbations. J Allergy Clin Immunol Pract. 2017; 5: 121–7.e2.
- 33. Marks GB, Dunn SM, Woolcock AJ. A scale for the measurement of quality of life in adults with asthma. J Clin Epidemiol. 1992;45:461-72.
- 34. American Thoracic Society, European Respiratory Society, ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide. Am J Respir Crit Care Med 2005. 2005;171:912–30.
- 35. Dweik RA, Boggs PB, Erzurum SC, Irvin CG, Leigh MW, Lundberg JO, Olin AC, Plummer AL, Taylor DR, American Thoracic Society Committee on Interpretation of Exhaled Nitric Oxide Levels for Clinical A. An official ATS clinical practice guideline: interpretation of exhaled nitric oxide levels (FENO) for clinical applications, Am J Respir Crit Care Med. 2011;184:602–15.
- 36. Oostveen E, MacLeod D, Lorino H, Farré R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003;22:1026-41.
- 37. Bonifazi M, Sverzellati N, Negri E, Pomponio G, Seletti V, Bonini M, Fraticelli P, Paolini L, Mattioli M, Franchi M, Tramacere I, Poletti V, La Vecchia C, Gasparini S, Gabrielli A. Increased prevalence of small airways dysfunction in patients with systemic sclerosis as determined by impulse oscillometry. Rheumatology (Oxford). 2019. pii:kez340.
- 38. Díaz Palacios MÁ, Hervás Marín D, Giner Valero A, Colomer Hernández N, Torán Barona C, Hernández Fernández de Rojas D. Correlation between

- impulse oscillometry parameters and asthma control in an adult population. J Asthma Allergy. 2019;12:195-203.
- 39. Chiu HY, Hsiao YH, Su KC, Lee YC, Ko HK, Perng DW. Small Airway Dysfunction by Impulse Oscillometry in Symptomatic Patients with Preserved Pulmonary Function. J Allergy Clin Immunol Pract. 2019. pii: S2213-2198(19)30608-7.
- 40. Beydon N, Davis SD, Lombardi E, Allen JL, Arets HG, Aurora P, Bisgaard H, Davis GM, Ducharme FM, Eigen H, Gappa M, Gaultier C, Gustafsson PM, Hall GL, Hantos Z, Healy MJ, Jones MH, Klug B, Lødrup Carlsen KC, McKenzie SA, Marchal F, Mayer OH, Merkus PJ, Morris MG, Oostveen E, Pillow JJ, Seddon PC, Silverman M, Sly PD, Stocks J, Tepper RS, Vilozni D, Wilson NM, American Thoracic Society/European Respiratory Society Working Group on Infant and Young Children Pulmonary Function Testing. An official American Thoracic Society/European Respiratory Society statement: pulmonary function testing in preschool children. Am J Respir Crit Care Med. 2007;175:1304-4.
- 41. Smith HJRP, Goldman MD. Forced oscillation technique and impulse oscillometry. Eur Respir Monogr. 2005;31:72–105.
- 42. Goldman MD. Clinical application of forced oscillation. Pulm Pharmacol Ther. 2001;14:341–50.
- 43. Nieto A, Pamies R, Oliver F, Medina A, Caballero L, Mazon A. Montelukast improves pulmonary function measured by impulse oscillometry in children with asthma (Mio study). Respir Med. 2006;100:1180–5.
- 44. Gonem S, Natarajan S, Desai D, Corkill S, Singapuri A, Bradding P, Gustafsson P, Costanza R, Kajekar R, Parmar H, Brightling CE, Siddiqui S. Clinical significance of small airway obstruction markers in patients with asthma. Clin Exp Allergy. 2014;44:499-507.
- 45. Lipworth B, Manoharan A, Anderson W. Unlocking the quiet zone: the small airway asthma phenotype. Lancet Respir Med. 2014;2:497-506.
- 46. Gourgoulianis K, Iliodromitis Z, Hatziefthimiou A, Molyvdas PA. Epithelium-dependent regulation of airways smooth muscle function. A histamine-nitric oxide pathway. Mediators Inflamm. 1998;7:409-11.
- 47. Gourgoulianis KI, Domali A, Molyvdas PA. Airway responsiveness: role of inflammation, epithelium damage and smooth muscle tension. Mediators Inflamm. 1999;8:261-3.
- 48. Andreou G, Karapetsas A, Gourgoulianis KI, Molyvdas PA. Left-handedness and inheritance of bronchial asthma. Percept Mot Skills. 2000;90:371-2.
- 49. Gourgoulianis K, Daniil Z, Athanasiou K, Rozou S, Bontozoglou V. Application of a One-Dimensional Computational Model for the Prediction of Deposition from a Dry Powder Inhaler. J Aerosol Med Pulm Drug Deliv. 2017;30:435-43.
- 50. Georgakakou S, GourgoulianisK, Daniil Z, Bontozoglou V. Prediction of particle deposition in the lungs based on simple modeling of alveolar mixing. Respir Physiol Neurobiol. 2016;225:8-18.

- 51. Gourgoulianis KI, Chatziparasidis G, Chatziefthimiou A, Molyvdas PA. Magnesium as a relaxing factor of airway smooth muscles. J Aerosol Med. 2001 Fall;14:301-7.
- 52. Kaditis AG, Gourgoulianis K, Winnie G. Anti-inflammatory treatment for recurrent wheezing in the first five years of life. Pediatr Pulmonol. 2003;35:241-52.
- 53. Krommydas G, Gourgoulianis KI, Andreou G, Kotrotsiou E, Raftopulos V, Paralikas T, Molyvdas PA. Fetal sensitivity to testosterone, left-handedness and development of bronchial asthma: a new approach. Med Hypotheses. 2004;62:143-5.
- 54. Kostikas K, Papaioannou AI, Tanou K, Koutsokera A, Papala M, Gourgoulianis KI. Portable exhaled nitric oxide as a screening tool for asthma in young adults during pollen season. Chest. 2008 Apr;133:906-13.
- 55. Koutsokera A, Loukides S, Gourgoulianis KI, Kostikas K. Biomarkers in the exhaled breath condensate of healthy adults: mapping the path towards reference values. Curr Med Chem. 2008;15:620-30.
- 56. Kostikas K, Koutsokera A, Papiris S, Gourgoulianis KI, Loukides S. Exhaled breath condensate in patients with asthma: implications for application in clinical practice. Clin Exp Allergy. 2008;38:557-65.
- 57. Oikonomidi S, Kostikas K, Tsilioni I, Tanou K, Gourgoulianis KI, Kiropoulos TS. Matrix metalloproteinases in respiratory diseases: from pathogenesis to potential clinical implications. Curr Med Chem. 2009;16:1214-28.
- 58. Zarogiannis S, Gourgoulianis KI, Kostikas K. Anti-interleukin-5 therapy and severe asthma. N Engl J Med. 2009 Jun 11;360(24):2576;
- 59. Papaioannou AI, Minas M, Tanou K, Gourgoulianis KI, Kostikas K. Exhaled NO may predict loss of asthma control: the effect of concomitant allergic rhinitis. Eur Respir J. 2009;34:1006-7.
- 60. Minas M, Papaioannou AI, Tsaroucha A, Daniil Z, Hatzoglou C, Sgantzos M, Gourgoulianis KI, Kostikas K. Body composition in severe refractory asthma: comparison with COPD patients and healthy smokers. PLoS One. 2010;5:e13233.
- 61. Malli F, Papaioannou Al, Gourgoulianis Kl, Daniil Z. The role of leptin in the respiratory system: an overview. Respir Res. 2010;11:152.
- 62. Kostikas K, Papaioannou AI, Tanou K, Giouleka P, Koutsokera A, Minas M, Papiris S, Gourgoulianis KI, Taylor DR, Loukides S. Exhaled NO and exhaled breath condensate pH in the evaluation of asthma control. Respir Med. 2011;105:526-32.
- 63. Zifa E, Daniil Z, Skoumi E, Stavrou M, Papadimitriou K, Terzenidou M, Kostikas K, Bagiatis V, Gourgoulianis KI, Mamuris Z. Mitochondrial genetic background plays a role in increasing risk to asthma. Mol Biol Rep. 2012;39:4697-708.

- 64. Stamatiou R, Paraskeva E, Gourgoulianis K, Molyvdas PA, Hatziefthimiou A. Cytokines and growth factors promote airway smooth muscle cell proliferation. ISRN Inflamm. 2012;2012:731472.
- 65. Tsaroucha A, Daniil Z, Malli F, Georgoulias P, Minas M, Kostikas K, Bargiota A, Zintzaras E, Gourgoulianis KI. Leptin, adiponectin, and ghrelin levels in female patients with asthma during stable and exacerbation periods. J Asthma. 2013;50:188-97.
- 66. Stamatiou R, Paraskeva E, Vasilaki A, Mylonis I, Molyvdas PA, Gourgoulianis K, Hatziefthimiou A. Long-term exposure to muscarinic agonists decreases expression of contractile proteins and responsiveness of rabbit tracheal smooth muscle cells. BMC Pulm Med. 2014;14:39.
- 67. Kotsiou OS, Gourgoulianis KI. Fractional exhaled nitric oxide: Signaling lung function changes in obstructive lung diseases. Ann Allergy Asthma Immunol. 2018;120:340.
- 68. Kotsiou OS, Peletidou S, Vavougios G, Karetsi E, Stavrou V, Zakynthinos G, Gourgoulianis KI, Daniil Z. Exhaled nitric oxide as a marker of chlorine exposure in young asthmatic swimmers. Ann Allergy Asthma Immunol. 2019;123:249-55.
- 69. Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry, Eur Respir J. 2005;26:319-38.
- 70. Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40:1324-43.
- 71. Millard RK. Key to better qualitative diagnostic calibrations in respiratory inductive plethysmography. Physiol Meas. 2002;23:N1–8.
- 72. Lo WLA, Huang DF. Assessment of an alternative calibration technique to record breathing pattern and its variability with respiratory inductive plethysmography. J Clin Monit Comput. 2017;31:755-64.